CLINICAL TRIAL: NCT04156438
Title: Early Use of Airway Pressure ReLease Ventilation in Critically Ill Adults With Moderate-to-severe Acute Respiratory Distress Syndrome
Brief Title: Airway Pressure Release Ventilation for Moderate-to-severe Acute Respiratory Distress Syndrome
Acronym: EARL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saskatchewan Health Authority - Regina Area (Other)
Responsible Party: Principal Investigator, Eric Sy, Critical Care Physician, Saskatchewan Health Authority - Regina Area
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB-19-51
Record Dates: First submitted 2019-10-26; First posted 2019-11-07 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Airway pressure release ventilation; low tidal volume ventilation; APRV; ARDSNet ventilation; LTVV; acute respiratory distress syndrome; ARDS
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low tidal volume ventilation (Active Comparator): Conventional low tidal volume ventilation
  Interventions: Device: Low tidal volume ventilation
- Airway pressure release ventilation (Experimental): Early use of airway pressure release ventilation
  Interventions: Device: Airway pressure release ventilation

INTERVENTIONS:
Device: Low tidal volume ventilation — Conventional ventilation strategy for patient with ARDS
  Arms: Low tidal volume ventilation
Device: Airway pressure release ventilation — Experimental ventilation protocol for patients with ARDS
  Arms: Airway pressure release ventilation

SUMMARY:
This study will examine the feasibility of a large clinical trial investigating the effectiveness of airway pressure release ventilation and low tidal volume ventilation for patients with moderate-to-severe acute respiratory distress syndrome.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) is a disease that has an incidence of 5% of hospitalized mechanically ventilated patients. ARDS is associated with high morbidity and mortality in critically ill patients, with mortality reported as high as 45% in severe ARDS. Patients who develop ARDS will require mechanical ventilation. Patients with ARDS are graded by the partial pressure of oxygen to fraction of inspired oxygen ratio (PaO2/FiO2) into three categories of severity: mild (PaO2/FiO2 201-300 mm Hg), moderate (PaO2/FiO2 101-200 mmHg), and severe (PaO2/FiO2 ≤ 100).

Volutrauma and barotrauma are thought to contribute to the development of ARDS and alter mortality. The damage that occurs to the lungs manifests itself as inflammation, which leads to poor gas exchange of oxygen and carbon dioxide. Several strategies of lung-protective mechanical ventilation have been investigated in ARDS, including the use of low tidal volume ventilation (LTVV) or ARDSNet strategy, high frequency oscillation ventilation (HFOV), and airway pressure release ventilation (APRV). Lung protective strategies may be best beneficial prior to the onset of the development of ARDS or early in the course of the disease. As a result of the ARDSNet trial, LTVV has been adopted as the usual standard of care of ventilation and safest mode of ventilation for patients with ARDS.

Recently, APRV has been proposed as a potential alternative to LTVV. APRV is a form of ventilation that keeps the lungs inflated through the majority of the breath cycle and allows patients to breathe spontaneously above this level of inflation. APRV allows for spontaneous respiration with increased airway pressure, potentially allowing for decreased sedation, shorter duration of mechanical ventilation, and decreased need for vasopressors. APRV has been associated with possible reduction in incidence of ARDS and in-hospital mortality in non-randomized observational studies. In patients with established ARDS, the use of APRV has also not been well studied, with most studies limited to small observational studies often with no comparison group. One randomized trial using APRV alone had less than 30% of patients having a diagnosis of ARDS and did not show any difference in any outcomes. Recently, Zhou and colleagues conducted a randomized trial comparing APRV to conventional ventilation in 138 mechanically ventilated patients with mild to severe ARDS and found that APRV may shorten the duration of mechanical ventilation and reduce intensive care unit (ICU) length of stay.

While some of these studies had shown promise of APRV compared to LTVV, there has not been acceptance of APRV into guidelines as first line ventilation, and recommendations of institutions such as the Canadian Agency for Drugs and Technology in Health (CADTH) recommends interpreting these results with caution. Consequently, there remains clinical equipoise on this issue. Some ICU clinicians will currently use APRV as a rescue mode of ventilation in ARDS in their clinical practice while others will continue with the use of LTVV. We would like to randomize patients to LTVV or APRV and examine the feasibility of conducting a large multicentre randomized controlled trial in Canada.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling the diagnostic criteria of ARDS, according to the Berlin definition
* Moderate to severe ARDS as defined as a PaO2: FiO2 ratio of ≤150 during invasive mechanical ventilation
* Endotracheal intubation and mechanical ventilation for ARDS less than 48 hours

Exclusion Criteria:

* Age less than 18 years
* Pregnancy
* Intracranial hypertension (suspected or confirmed)
* Severe chronic obstructive pulmonary disease as defined by either:

  1. FEV1/FVC less than 50% predicted, or
  2. Chronic hypercarbia (PaCO2>45 mmHg), chronic hypoxemia (PaO2 < 55 mmHg) on room air, and/or elevated admission serum HCO3 >30 mmol/L
* Presence of documented barotrauma, i.e. pneumothorax
* Treatment with extracorporeal support (ECMO) at enrollment
* Refractory shock
* Advanced directives indicating preferences to not have advanced life support
* Moribund patient, i.e. not expected to survive longer than 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Informed consent rate | Informed consent rate will be measured over a 1 year period of the pilot study
  A successful informed consent rate will be defined as ≥70% of substitute decision makers or patients approached choosing to participate in this trial
Recruitment rate | Recruitment rate will be measured over the one year of the pilot study.
  A successful recruitment rate will be achieving at least 15 patients over the 1 year period.
Protocol adherence rate | Protocol adherence will be measured for each study patient, and compiled over the duration of the pilot study (i.e. 1 year).
  An adherence rate of at least 80% will be considered successful.

SECONDARY OUTCOMES:
28-day mortality | Up to Day 28
  Death, measured from time of enrollment until 28 days.
In-hospital mortality | Up to 365 days
  Death, at hospital discharge
ICU length of stay | Up to 365 days
  Length of stay in the intensive care unit
Hospital length of stay | Up to 365 days
  Length of stay in the hospital in days
Length/duration of mechanical ventilation | Up to 365 days
  Length of time patient was on mechanical ventilation
Incidence of tracheostomy | Up to 365 days
  Incidence of tracheostomy during their ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Sy, MD MPH FRCPC, Principal Investigator — Saskatchewan Health Authority - Regina Area
Locations (1):
- Regina General Hospital, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Walkey AJ, Summer R, Ho V, Alkana P. Acute respiratory distress syndrome: epidemiology and management approaches. Clin Epidemiol. 2012;4:159-69. doi: 10.2147/CLEP.S28800. Epub 2012 Jul 16. PMID 22866017
- [Background] Gattinoni L, Pesenti A. The concept of "baby lung". Intensive Care Med. 2005 Jun;31(6):776-84. doi: 10.1007/s00134-005-2627-z. Epub 2005 Apr 6. PMID 15812622
- [Background] de Haro C, Martin-Loeches I, Torrents E, Artigas A. Acute respiratory distress syndrome: prevention and early recognition. Ann Intensive Care. 2013 Apr 24;3(1):11. doi: 10.1186/2110-5820-3-11. PMID 23617961
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Ferguson ND, Cook DJ, Guyatt GH, Mehta S, Hand L, Austin P, Zhou Q, Matte A, Walter SD, Lamontagne F, Granton JT, Arabi YM, Arroliga AC, Stewart TE, Slutsky AS, Meade MO; OSCILLATE Trial Investigators; Canadian Critical Care Trials Group. High-frequency oscillation in early acute respiratory distress syndrome. N Engl J Med. 2013 Feb 28;368(9):795-805. doi: 10.1056/NEJMoa1215554. Epub 2013 Jan 22. PMID 23339639
- [Background] Young D, Lamb SE, Shah S, MacKenzie I, Tunnicliffe W, Lall R, Rowan K, Cuthbertson BH; OSCAR Study Group. High-frequency oscillation for acute respiratory distress syndrome. N Engl J Med. 2013 Feb 28;368(9):806-13. doi: 10.1056/NEJMoa1215716. Epub 2013 Jan 22. PMID 23339638
- [Background] Jain SV, Kollisch-Singule M, Sadowitz B, Dombert L, Satalin J, Andrews P, Gatto LA, Nieman GF, Habashi NM. The 30-year evolution of airway pressure release ventilation (APRV). Intensive Care Med Exp. 2016 Dec;4(1):11. doi: 10.1186/s40635-016-0085-2. Epub 2016 May 20. PMID 27207149
- [Background] Andrews PL, Shiber JR, Jaruga-Killeen E, Roy S, Sadowitz B, O'Toole RV, Gatto LA, Nieman GF, Scalea T, Habashi NM. Early application of airway pressure release ventilation may reduce mortality in high-risk trauma patients: a systematic review of observational trauma ARDS literature. J Trauma Acute Care Surg. 2013 Oct;75(4):635-41. doi: 10.1097/TA.0b013e31829d3504. PMID 24064877
- [Background] Futier E, Constantin JM, Paugam-Burtz C, Pascal J, Eurin M, Neuschwander A, Marret E, Beaussier M, Gutton C, Lefrant JY, Allaouchiche B, Verzilli D, Leone M, De Jong A, Bazin JE, Pereira B, Jaber S; IMPROVE Study Group. A trial of intraoperative low-tidal-volume ventilation in abdominal surgery. N Engl J Med. 2013 Aug 1;369(5):428-37. doi: 10.1056/NEJMoa1301082. PMID 23902482
- [Background] Serpa Neto A, Cardoso SO, Manetta JA, Pereira VG, Esposito DC, Pasqualucci Mde O, Damasceno MC, Schultz MJ. Association between use of lung-protective ventilation with lower tidal volumes and clinical outcomes among patients without acute respiratory distress syndrome: a meta-analysis. JAMA. 2012 Oct 24;308(16):1651-9. doi: 10.1001/jama.2012.13730. PMID 23093163
- [Background] Maxwell RA, Green JM, Waldrop J, Dart BW, Smith PW, Brooks D, Lewis PL, Barker DE. A randomized prospective trial of airway pressure release ventilation and low tidal volume ventilation in adult trauma patients with acute respiratory failure. J Trauma. 2010 Sep;69(3):501-10; discussion 511. doi: 10.1097/TA.0b013e3181e75961. PMID 20838119
- [Background] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Background] Habashi NM. Other approaches to open-lung ventilation: airway pressure release ventilation. Crit Care Med. 2005 Mar;33(3 Suppl):S228-40. doi: 10.1097/01.ccm.0000155920.11893.37. PMID 15753733
- [Background] Lim J, Litton E, Robinson H, Das Gupta M. Characteristics and outcomes of patients treated with airway pressure release ventilation for acute respiratory distress syndrome: A retrospective observational study. J Crit Care. 2016 Aug;34:154-9. doi: 10.1016/j.jcrc.2016.03.002. Epub 2016 Mar 9. PMID 27020770
- [Background] Sydow M, Burchardi H, Ephraim E, Zielmann S, Crozier TA. Long-term effects of two different ventilatory modes on oxygenation in acute lung injury. Comparison of airway pressure release ventilation and volume-controlled inverse ratio ventilation. Am J Respir Crit Care Med. 1994 Jun;149(6):1550-6. doi: 10.1164/ajrccm.149.6.8004312.
- [Background] Zhou Y, Jin X, Lv Y, Wang P, Yang Y, Liang G, Wang B, Kang Y. Early application of airway pressure release ventilation may reduce the duration of mechanical ventilation in acute respiratory distress syndrome. Intensive Care Med. 2017 Nov;43(11):1648-1659. doi: 10.1007/s00134-017-4912-z. Epub 2017 Sep 22. PMID 28936695
- [Background] Seal K, Featherstone R. Airway Pressure Release Ventilation for Acute Respiratory Distress Syndrome: Clinical Effectiveness and Guidelines [Internet]. Ottawa (ON): Canadian Agency for Drugs and Technologies in Health; 2018 Feb 1. Available from http://www.ncbi.nlm.nih.gov/books/NBK531787/ PMID 30307725